CLINICAL TRIAL: NCT02269904
Title: Fluorouracil Implants（SinoFuan®）Used for Intraperitoneal Chemotherapy During Operation for Intraperitoneal Chemotherapy During Operation for Treatment of Phase III Gastric Cancer, Randomized, Controlled, Multicentres Open Study.
Brief Title: Fluorouracil Implants Used for Intraperitoneal Chemotherapy During Operation for Treatment of Phase III Gastric Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sinofuan01
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: DSF

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluorouracil Implants and Xelox regimes (Active Comparator): Fluorouracil Implants: 800mg, implanted in the abdominal cavity during operation.
  Xelox regimes: Capecitabine,1000 mg/m2，PO.BID, from D1 to D14; Oxaliplatin, 130 mg/m2，IV, D1 in each cycle. The cycle will repeated every 21 days till 6 cycles finished.
  Interventions: Drug: Fluorouracil Implants; Drug: Xelox regimes
- Xelox regimes (Active Comparator): Xelox regimes: Capecitabine,1000 mg/m2，PO.BID, from D1 to D14; Oxaliplatin, 130 mg/m2，IV, D1 in each cycle. The cycle will repeated every 21 days till 6 cycles finished.
  Interventions: Drug: Xelox regimes

INTERVENTIONS:
Drug: Fluorouracil Implants — Fluorouracil Implants: 800mg, implanted in the abdominal cavity during operation.
  Arms: Fluorouracil Implants and Xelox regimes
Drug: Xelox regimes — Xelox regimes: Capecitabine,1000 mg/m2，PO.BID, from D1 to D14; Oxaliplatin, 130 mg/m2，IV, D1 in each cycle. The cycle will repeated every 21 days till 6 cycles finished.

SUMMARY:
SinoFuan is a kind of Fluorouracil Implants for intraperitoneal chemotherapy during operation for treatment of gastric cancer. The indication has bee approved by Chinese FDA. The study is a post-marketing study. The subjects will be divided into two groups (Group A and Group B ). The subject in Group A will receive D2 radical gastrectomy(R0),Sinofuan during operation and 6 cycles of Xelox adjuvant chemotherapy.The subject in Group B will receive D2 radical gastrectomy(R0),and 6 cycles of Xelox adjuvant chemotherapy. The subject's benefits from SinoFuan will be analyzed through comparing 3 years DFS of two groups.

ELIGIBILITY:
Inclusion Criteria:

1. primary gastric cancer, Phase III
2. D2 radical gastrectomy(R0)
3. 18 year old or above
4. KPS≥70%；
5. suitable hematologic function: ANC≥1.5×109/L, PLC≥80×109/L
6. suitable liver function: Total bilirubin≤1.5×normal ULN, AST and ALT≤2.5×normal ULN.
7. suitable renal function: Cr≤1.5×normal ULN,or Ccr≥50 ml/min 8 .for the female subject, pregnancy test must be negative in 27 hours before enrollment .

9. the authorized ICF must be signed

Exclusion Criteria:

1. non-initial gastric cancer；
2. having the other uncontrolled diseases.
3. obvious loss of weight ( more than 10% within 6 weeks )
4. the female in pregnancy or feeding.
5. contraindication to study drug
6. participating in other clinical trial and at the time of treatment period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
DFS (Disease Free Survival) | 3 year
  During 3 years of monitoring period, any cancer relapse will be recorded

SECONDARY OUTCOMES:
adverse event | 3 years
  During 3 years of monitoring period, any AEs will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Heilongjiang Cancer Hospital, Harebin, Heilongjiang, China

REFERENCES:
- [Derived] Xu Y, Zhang R, Li C, Sun Z, Deng J, Wang X, Ding X, Wang B, Xue Q, Ke B, Zhan H, Liu N, Liu Y, Wang X, Liang H, Xue Y, Xu H. Intraperitoneal Chemotherapy Using Fluorouracil Implants Combined With Radical Resection and Postoperative Adjuvant Chemotherapy for Stage III Gastric Cancer: A Multi-Center, Randomized, Open-Label, Controlled Clinical Study. Front Oncol. 2021 Jul 8;11:670651. doi: 10.3389/fonc.2021.670651. eCollection 2021. PMID 34307140